CLINICAL TRIAL: NCT05177978
Title: The Chronic Cognitive Effects of 6- and 12-weeks Administration of a Food Supplement Containing Phosphatidylserine: A Double Blind, Randomized, Placebo Controlled, Parallel Groups Study in Healthy Children Aged 8 to 12 Years
Brief Title: The Cognitive Effects of 6- and 12-weeks Administration of a Food Supplement Containing Phosphatidylserine in Healthy Children Aged 8 to 12 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: International Flavors & Fragrances Inc. (Unknown)
Responsible Party: Principal Investigator, Philippa Jackson, Principal Investigator, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 39BZ1
Record Dates: First submitted 2021-08-04; First posted 2022-01-05 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Cognitive Change
Keywords: Cognition; Phosphatidylserine; Memory; Learning; Attention
MeSH Terms: interventions — Phosphatidylserines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phosphatidylserine (Experimental): 100 mg elemental phosphatidylserine
  Interventions: Dietary Supplement: Phosphatidylserine
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phosphatidylserine — Phosphatidylserine containing supplement (2 x chewable gummies/day; Total daily dose of 100 mg elemental phosphatidylserine)
  Arms: Phosphatidylserine
Dietary Supplement: Placebo — Placebo comparator (2 x chewable gummies/day, matched to shape and color without active ingredient)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the cognitive effects (attention, learning, and memory) of 6 and 12 weeks administration of a supplement containing phosphatidylserine in comparison to a placebo in healthy children aged 8 to 12 years old. The study will utilize Rey Auditory Verbal Learning Test (RAVLT) and Computerised Mental Performance Assessment System (COMPASS, Northumbria University) for a broad assessment of cognitive function/learning, and actigraphy to monitor sleep.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be in good health as reported by themselves and their parent/guardian.
* Healthy children aged 8 to 12 years and enrolled in school years 4 to 7 at the time of giving consent
* Have been speaking English at school since reception
* Willingness of the children and parents to give their written informed consent, according to GCP and local regulations and being able to participate in all scheduled visits, intervention plans, tests and other trial procedures
* Children with a normal sex and age-related BMI according to the local NHS guidelines (3rd to 90th percentiles)

Exclusion Criteria:

* Relevant allergy or known hypersensitivity to one of the ingredients contained in the investigational drug.
* Are currently taking any illicit, herbal or recreational drugs including alcohol and tobacco.
* Taking any prescribed or OTC medication against chronic or non- chronic illnesses.
* Have used dietary supplements within the last 4 weeks
* Are diagnosed with ADHD, dyslexia or any neurodevelopmental disorder or learning difficulty.
* Suffer from visual (including colour blindness) or hearing impairment (that may impact task performance in the opinion of the PI.
* Have any serious illness, cognitive impairment or medical disorder that may confound with study results or interfere with compliance.
* Have any other active or unstable medical condition, that, in the opinion of the PI, may adversely affect the participant's ability to complete the study
* Are experiencing exceptional social/family stressors.
* Consume more than one portion (>100g) per week of the following dietary sources high in phosphatidylserine: Oily fish such as salmon, mackerel, herring, tuna and eel. Animal internal organs such as liver, kidney, brain and heart. Note: Information on continued adherence to this criteria will be captured within treatment diary. If a child continuously consumes more than one portion per week of PS rich food the sponsor will be informed on a case by case basis. If deemed to be significant, they will be excluded, (but allowed to continue the study to the end (day 84)) and will be replaced.
* Subjects that have followed specific diet, e.g. high protein diet, within 30 days prior to study start
* Serious diet change, e.g. Ketogenic or vegan, within 30 days prior to study start.
* Consumption of > 250 mg/day of caffeine.
* Are unable to complete all of the study assessments
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 8 weeks
* Are non-compliant with regards treatment consumption

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
COMPASS global performance measures | Following 12 weeks of intervention
  Speed of performance, and accuracy of performance measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Cognitive domain factor score | Following 12 weeks of intervention
  Speed of attention, accuracy of attention, speed of memory, accuracy of working memory, and accuracy of episodic memory measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Location Learning score | Following 12 weeks of intervention
  Learning index, displacement score, and delayed recall score, measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Rey Auditory Verbal Learning Test (RAVLT) | Following 12 weeks of intervention
  Learning score, Immediate recall, delayed recall, and delayed recognition measured by the Rey Auditory Verbal Learning Test

SECONDARY OUTCOMES:
COMPASS global performance measures | Following 6 weeks of intervention
  Speed of performance, and accuracy of performance measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Cognitive domain factor score | Following 6 weeks of intervention
  Speed of attention, accuracy of attention, speed of memory, accuracy of working memory, and accuracy of episodic memory measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Location Learning score | Following 6 weeks of intervention
  Learning index, displacement score, and delayed recall score, measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Rey Auditory Verbal Learning Test (RAVLT) | Following 6 weeks of intervention
  Learning score, Immediate recall, delayed recall, and delayed recognition measured by the Rey Auditory Verbal Learning Test
Individual cognitive task score | Following 6 and 12 weeks of intervention
  Individual tasks include the following: immediate word recall, simple reaction time, choice reaction time, 4 choice reaction time, arrows flankers, digit vigilance, rapid visual information processing, Stroop, Corsi blocks, numeric working memory, 2-back, delayed word recall, delayed picture recognition, and delayed word recognition measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Children's Sleep Habits Questionnaire (CSHQ) | Following 6 and 12 weeks of intervention
  23 items questionnaire completed by the parent, with a 3-point scale where a higher score is indicative of more disturbed sleep.
Children's Sleep self-report (SSR) questionnaire | Following 6 and 12 weeks of intervention
  26 items questionnaire completed by the child with a 3-point scale where a higher score is indicative of more disturbed sleep.
Sleep measures | Following 12 weeks of intervention
  Sleep actigraphy device (measuring: sleep onset, total sleep time (TST), wake after sleep onset (WASO), awakenings, average awakening, efficiency) and sleep duration as reported in a sleep diary.
Parent Visual Analogue Scales (VAS) | Following 6 and 12 weeks of intervention
  100 mm VAS in which the parent rates their child via the following parameters: Attention, performance at school, performance of schoolwork at home, happiness, and stress.
Child mood Visual Analogue Scales (VAS) | Following 6 and 12 weeks of intervention
  100 mm VAS questionnaire in which the child rates their own mood via the following parameters: Relaxed, alert, jittery, tense, tired, headache, overall mood, mental fatigue, performance, happy/sad, and stress /calm

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Jackson, Principal Investigator — Northumbria University
Locations (1):
- Brain, Performance, Nutrition Research Centre, Northumbria University, Newcastle upon Tyne, Tyne & Wear, United Kingdom

REFERENCES:
- [Derived] Friling M, Jackson PA, Kennedy D, Dodd F, Smith E, Lavie A, Lopresti A, Ivanir E, Jalanka J. The cognitive effects of supplementation with sunflower phosphatidyl serine in healthy children aged 8 to 12 years: a randomized controlled trial. Nutr J. 2025 Nov 29;25(1):3. doi: 10.1186/s12937-025-01264-9. PMID 41318468